CLINICAL TRIAL: NCT05189912
Title: Clinical Study on the Application of a Specimen Retrieving Bag in Endoscopic Polypectomy to Reduce the Polyp Fragmentation Rate
Brief Title: Clinical Study on the Application of a Specimen Retrieving Bag to Reduce the Polyp Fragmentation Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Polyp bag frag
Record Dates: First submitted 2021-12-28; First posted 2022-01-13 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Colonic Polyp
Keywords: Colonic Polyp; Specimen retrieval bag; Polyp fragmentation
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients were not informed about their randomization allocation in order to increase reliability during follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specimen retrieving bag group (Experimental): Resected polyps were retrieved by specimen retrieving bag. This group was set as a experimental group.
  Interventions: Device: Specimen retrieving bag
- Suction group (Active Comparator): Resected polyps were retrieved by removing the colonoscope suction valve and connecting a polyp trap to suction onto the instrument channel port.
  This group was set as a control group.
  Interventions: Behavioral: Sucking polyps to the instrument channel port

INTERVENTIONS:
Device: Specimen retrieving bag — Specimen retrieving bag was used to retrieve resected polyps.
  Arms: Specimen retrieving bag group
Behavioral: Sucking polyps to the instrument channel port — Remove the colonoscope suction valve and connect a polyp trap to suction onto the instrument channel port.
  Arms: Suction group

SUMMARY:
It is necessary to retrieve the resected polyp to determine the pathological nature of polyp and to judge the completeness of resection in polypectomy. For polyps with a larger diameter (>5mm), the most reliable way to retrieve them is to suck them out with the colonoscope. However, this method requires multiple colonoscope insertions, resulting in prolonged operation time and increased patient suffering. Therefore, clinicians often receive polyps by pressing the colonoscope suction valve. But it is difficult to receive polyps or even fail to receive. Even if the polyps were successfully received by this method, many polyps were fragmented. When the polyp is fragmented, the pathologist cannot be sure of the completeness of the polyp removal.

By removing the colonoscope suction valve and connecting a polyp trap to suction onto the instrument channel port, the polyp fragmentation rate was reduced greatly. To further reduce the polyp fragmentation rate, while reducing the operation time and colon insertions, we applied the polyp receiving bag in colonoscopy operations. The primary purpose of this study is to evaluate the effectiveness of the application of the polyp retrieving bag to reduce the polyp fragmentation rate.

DETAILED DESCRIPTION:
After polyp resection, it is necessary to retrieve the resected polyp to determine the pathological nature of polyp and to judge the completeness of resection in polypectomy. For polyps with a small diameter (≤5mm), usually by pressing the suction valve button of the colonoscope, polyps could be completely retrieved through a trap. For polyps with a larger diameter (>5mm), the most reliable way to retrieve them is to suck them out with the colonoscope. However, this method requires multiple colonoscope insertions, resulting in prolonged operation time and increased patient suffering. Therefore, clinicians often receive resected polyps with larger diameters by pressing the colonoscope suction valve. However, it is difficult to receive polyps or even fail to receive. Even if the polyps were successfully received, many polyps were fragmented, and the polyp fragmentation rate can be as high as 36.6%~ 60.3%. When the polyp is fragmented, the pathologist cannot be sure of the completeness of the polyp removal. Due to the possibility of malignant transformation in some polyps, the completeness of polyp resection is essential to guide the following treatment.

Some effective methods were developed to reduce polyp fragmentation, including removing the colonoscope suction valve and connecting a polyp trap to suction onto the instrument channel port. The resulting polyp fragmentation rates are 22.4-43.0% and 18.5%, respectively. To further reduce the polyp fragmentation rate, while reducing the operation time and improving the efficiency of the operation, we applied the polyp receiving bag in colonoscopy operations. In a previous pilot study, the polyp receiving bag has been applied in clinical practice, and its polyp fragmentation rate and polyp recovery failure rate are quite low. The primary purpose of this study is to evaluate the effectiveness of the application of the Polyp retrieving bag to reduce the polyp fragmentation rate.

ELIGIBILITY:
Inclusion Criteria:

1. Single polyp, with a diameter of 5-15mm,
2. Written informed consent.

Exclusion Criteria:

1. Polyps that were not removed en bloc,
2. Underlying bleeding disorder,
3. The platelet count less than 50×10^9/L,
4. Serious cardio-pulmonary, hepatic or renal disease,
5. Intolerance to endoscopy,
6. Other high-risk conditions or disease (such as massive ascites, etc.),
7. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-14 (Actual)

PRIMARY OUTCOMES:
Polyp fragmentation rate | 1 day
  The proportion of fragmented polyps to all polyps.

SECONDARY OUTCOMES:
Retrieving failure rate | 1 day
  The proportion of polyps that failed to be retrieved to all polyps removed.
The duration time of polyp resection | 1day
  The duration time of polyp resection to the colonoscopy withdraw from body.
The insertion times of colonoscopy | 1 day
  The insertion times of colonoscopy during the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, MD, Principal Investigator — Beijing 302 Hospital
Locations (1):
- The Fifth Medical Center of Chinese PLA General Hosptial, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chu J, Ma C, Min M, Bi Q, Shen W, Zhang X, Zhang H, Li A, Liu Y, Lu Z. A novel polyp retrieval bag reduces the polyp fragmentation rate in colon polypectomy: a single-blind randomized controlled study. Int J Colorectal Dis. 2024 Jul 24;39(1):118. doi: 10.1007/s00384-024-04694-9. PMID 39048748